CLINICAL TRIAL: NCT05786391
Title: Trendelenburg, Abdominal Insufflation and Time to Completion of Cystoscopy A Prospective Randomized Trial
Brief Title: Trendelenburg, Abdominal Insufflation and Time to Completion of Cystoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Randa Jalloul, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSC-MS-22-1081
Record Dates: First submitted 2023-03-05; First posted 2023-03-27 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Bladder Integrity; Bladder Function; Ureteral Integrity; Ureteral Function
MeSH Terms: interventions — Head-Down Tilt; Insufflation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Flat position with no Insufflation (Experimental)
  Interventions: Other: Flat position
- Trendelenburg position and Insufflation (Experimental): insufflation to 15 mm Hg
  Interventions: Other: Trendelenburg position; Device: Insufflation
- Flat position and Insufflation (Experimental)
  Interventions: Other: Flat position; Device: Insufflation
- Trendelenburg position with no Insufflation (Experimental)
  Interventions: Other: Trendelenburg position

INTERVENTIONS:
Other: Flat position — Flat patient position during the cystoscopy
  Arms: Flat position and Insufflation; Flat position with no Insufflation
Other: Trendelenburg position — Trendelenburg position (head down) during the cystoscopy
  Arms: Trendelenburg position and Insufflation; Trendelenburg position with no Insufflation
Device: Insufflation — Insufflation to 15 mm Hg
  Arms: Flat position and Insufflation; Trendelenburg position and Insufflation

SUMMARY:
Objective:

The investigators seek to compare the efficiency of the cystoscopy with two interventions:

1. patient position during the cystoscopy (Trendelenburg (head down) or flat)
2. Abdominal insufflation (insufflation versus no insufflation)

DETAILED DESCRIPTION:
This is a randomized controlled trial assessing time to completion of cystoscopy in seconds after minimally invasive gynecologic surgery.

The investigators seek to compare the efficiency of the cystoscopy with two interventions:

1. patient position during the cystoscopy (Trendelenburg (head down) or flat)
2. Abdominal insufflation (insufflation versus no insufflation).

Both interventions are used as usual care and depend on surgeon preference without evidence why one would be faster at completing the cystoscopy. Also note that these two interventions are performed multiple times during the surgery itself and outside the cystoscopy procedure routinely. The investigator's main objective is to assess which intervention or combination of interventions is more efficient.

ELIGIBILITY:
Inclusion Criteria:

- Patient undergoing Planned cystoscopy in the benign gynecology service, (specifically undergoing a laparoscopic or robotic procedure requiring insufflation).

Exclusion Criteria:

* Pregnancy
* Known urologic anomaly
* Unplanned cystoscopy
* Cancer surgery
* Urogynecology surgery
* comorbidities including cardiac disease, chronic hypertension, any stage kidney disease (including abnormal creatinine level), and use of diuretics.
* Undergoing extensive ureterolysis
* Blood loss more than 500 milliliters (mLs)
* Contra-indications to position change and insufflation

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randa Jalloul, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flat Position With no Insufflation | Trendelenburg Position and Insufflation | Flat Position and Insufflation | Trendelenburg Position With no Insufflation
Started | 31 | 30 | 30 | 31
Completed | 31 | 30 | 30 | 31
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flat Position With no Insufflation | Trendelenburg Position and Insufflation | Flat Position and Insufflation | Trendelenburg Position With no Insufflation | Total
Number analyzed (Participants) | 31 | 30 | 30 | 31 | 122
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 45 [41 to 48] | 44 [41 to 48] | 46 [42 to 49] | 45 [42 to 51] | 45 [41 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 30 | 31 | 122
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 9 | 6 | 7 | 6 | 28
  Other (non-Caucasian) | 22 | 24 | 23 | 25 | 94
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 30 | 31 | 122
Number of participants with Diabetes [Count of Participants; unit: Participants] | 3 | 3 | 3 | 4 | 13
Number of participants with hypertension [Count of Participants; unit: Participants] | 9 | 9 | 1 | 10 | 29
Number of participants who smoke [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0 | 0
Number of participants with hyperlipidemia [Count of Participants; unit: Participants] | 1 | 6 | 2 | 4 | 13
Number of participants with heart disease [Count of Participants; unit: Participants] | 1 | 0 | 1 | 2 | 4
Number of participants with lung disease [Count of Participants; unit: Participants] | 0 | 2 | 2 | 2 | 6
Number of Participants with history of previous abdominal surgery [Count of Participants; unit: Participants] | 17 | 26 | 20 | 21 | 84
Parity [Count of Participants; unit: Participants] — number of completed pregnancies beyond 20 weeks gestation (whether viable or nonviable)
  Participants
    0 | 26 | 26 | 27 | 22 | 101
    1 or more | 5 | 4 | 3 | 9 | 21
Level of Creatinine [Median (Inter-Quartile Range); unit: milligrams per deciliter] — Population: Data were not collected for 1 participant in the Trendelenburg position and Insufflation arm.
  milligrams per deciliter
    number analyzed (Participants) | 31 | 29 | 30 | 31 | 121
    (all) | 0.78 [0.71 to 0.84] | 0.78 [0.70 to 0.91] | 0.71 [0.57 to 0.83] | 0.82 [0.75 to 0.94] | 0.78 [0.68 to 0.86]
Hemoglobin level at admission [Median (Inter-Quartile Range); unit: grams per deciliter] | 12.40 [10.95 to 13.25] | 12.05 [10.90 to 13.38] | 11.45 [9.63 to 12.85] | 12.00 [11.05 to 12.90] | 12.00 [10.60 to 13.10]
Hemoglobin A1c (HbA1c) at Pre-operation [Median (Inter-Quartile Range); unit: percentage of HbA1c] — Population: Data were not collected for 25 participants in the Flat position with no Insufflation arm. Data were not collected for 25 participants in the Trendelenburg position and Insufflation arm. Data were not collected for 25 participants in the Flat position and Insufflation arm. Data were not collected for 23 participants in the Trendelenburg position with no Insufflation arm.
  percentage of HbA1c
    number analyzed (Participants) | 6 | 5 | 5 | 8 | 24
    (all) | 5.35 [5.13 to 5.58] | 5.80 [5.60 to 6.00] | 5.50 [5.40 to 5.60] | 6.00 [5.60 to 6.40] | 5.60 [5.30 to 6.05]
Glomerular Filtration Rate (GFR) at admission [Median (Inter-Quartile Range); unit: milliliters per minutes] — Population: Data were not collected for 1 participant in the Trendelenburg position and Insufflation arm.
  milliliters per minutes
    number analyzed (Participants) | 31 | 29 | 30 | 31 | 121
    (all) | 96 [88 to 107] | 94 [82 to 108] | 106 [88 to 114] | 88 [76 to 101] | 96 [82 to 108]
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 30 [26 to 35] | 31 [28 to 34] | 31 [25 to 37] | 35 [28 to 42] | 31 [26 to 36]

OUTCOME MEASURES:

1. Primary Outcome: Time in Seconds to Complete the Cystourethroscopy
Description: Time in seconds to satisfactorily complete the cystourethroscopy (including visualization of the dome, the ureteral jets, the bladder mucosa, and the urethra).
Time Frame: From the start of the cystoscopy to the completion of the cystoscopy (about 4 minutes)
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Flat Position With no Insufflation | Trendelenburg Position and Insufflation | Flat Position and Insufflation | Trendelenburg Position With no Insufflation
Number analyzed (Participants) | 31 | 30 | 30 | 31
seconds | 103 [65 to 184] | 117 [50 to 223] | 147 [71 to 208] | 82 [71 to 136]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Flat Position With no Insufflation | Trendelenburg Position and Insufflation | Flat Position and Insufflation | Trendelenburg Position With no Insufflation
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 1/31 | 2/30 | 1/30 | 0/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flat Position With no Insufflation (N=31) | Trendelenburg Position and Insufflation (N=30) | Flat Position and Insufflation (N=30) | Trendelenburg Position With no Insufflation (N=31)
Dizziness (General disorders) | 0 | 0 | 1 | 0 — Adverse event is not related to intervention.
Fall (General disorders) | 0 | 1 | 0 | 0 — Adverse event is not related to intervention.
Post-Operation abdominal pain (General disorders) | 0 | 1 | 0 | 0 — Adverse event is not related to intervention.
Vaginal Bleeding (General disorders) | 1 | 0 | 0 | 0 — Adverse event is not related to intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT05786391/Prot_SAP_000.pdf